CLINICAL TRIAL: NCT04619238
Title: Reliability of The King's Health Questionnaire and the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form in Assessing Urinary Incontinence Effects in Polish Women
Brief Title: Reliability of KHQ and ICIQ-SF in Assessing Urinary Incontinence Effects in Polish Women
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Katarzyna Skorupska, Principal investigator, Medical University of Lublin
Other Study IDs: 2\2020
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Urinary Incontinence; Overactive Bladder; Stress Urinary Incontinence; Urge Incontinence
Keywords: king's health questionnaire; the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- no urinary incontinence: patients without UI
  Interventions: Diagnostic Test: King's Health Questionnaire; Diagnostic Test: the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form
- stress urinary incontinence: patients with SUI
  Interventions: Diagnostic Test: King's Health Questionnaire; Diagnostic Test: the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form
- overactive bladder: patients with OAB
  Interventions: Diagnostic Test: King's Health Questionnaire; Diagnostic Test: the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form
- mix urinary incontinence: patients with MUI
  Interventions: Diagnostic Test: King's Health Questionnaire; Diagnostic Test: the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form
- Urge: patients with urge incontinence
  Interventions: Diagnostic Test: King's Health Questionnaire; Diagnostic Test: the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form

INTERVENTIONS:
Diagnostic Test: King's Health Questionnaire — patients fulfilled questionnaire
Diagnostic Test: the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form — patients fulfilled ICIQ-SF questionnaire

SUMMARY:
The aim of this study was to assess the psychometric properties of KHQ and ICIQ-SF in polish women.

DETAILED DESCRIPTION:
Purpose The King's Health Questionnaire (KHQ) and the International Consultation on Incontinence Modular Questionnaire (ICIQ-SF) Short Form are widely used in clinical practice. The aim of this study was to assess the psychometric properties of KHQ and ICIQ-SF in polish women.

Methods One hundred fifty-five women with urinary incontinence (UI) aged between 19-82 years underwent urodynamic investigation and completed both KHQ and ICIQ-SF. To evaluate the factor structure and construct the validity of the KHQ and ICIQ, Principal Component Analysis (PCA) using VARIMAX rotation was conducted for all questionnaire items. PCA results were also confirmed by Spearman's correlations between KHQ and ICIQ items. Moreover, the internal consistency of the KHQ and ICIQ was estimated by way of Cronbach's alpha coefficient (α). Statistical analysis was performed using STATISTICA version 13.1 software (StatSoft, Poland), as well as open source R software (version 3.4.4).

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patients with symptoms of urinary incontinence
* age 18-82 years

Exclusion Criteria:

* lack of consent
* inability to understand the study protocol

Ages: 18 Years to 82 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women age 18-82 years who declared symptoms of urinary incontinence
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
psychometric properties of KHQ in polish women with urinary incontinence | 2017-2018
  psychometric properties of KHQ
psychometric properties of ICIQ-SF in polish women with urinary incontinence | 2017-2018
  psychometric properties of ICIQ-SF

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Rechberger, Professor, Study Director — Medical University of Lublin
Locations (1):
- Katarzyna Skorupska, Lublin, Poland